CLINICAL TRIAL: NCT00566059
Title: Comparison Between Invasive Coronary Angiography and Dual-Source Computed Tomography
Brief Title: Computed Tomographic Angiography or Conventional Coronary Angiography in Clinical Decision Making
Acronym: CARDUCCI
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: F. Zijlstra, University Medical Center Groningen
Other Study IDs: CARDUCCI
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis
Keywords: therapeutic advice
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients planned for elective conventional coronary angiography will undergo CT coronary angiography (Dual Source CT) in order to assess the correlation of stenosis detection and therapeutic advice between conventional and CT coronary angiography. We hypothesize that their is a good correlation between conventional and CT coronary angiography for stenosis detection and therapeutic advice.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age
* Scheduled for elective coronary angiography

Exclusion Criteria:

* Patients with known iodine allergy
* Severe renal insufficiency (creatinine levels > 120 micromol/L)
* Hyperthyroidism
* Cardiac arrhythmias
* Unstable clinical condition
* Inability to follow breath-hold commands
* Previous PCI or CABG were excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 50 years of age, scheduled for elective coronary angiography
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-05; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Zijlstra, MD PhD, Study Director — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands